CLINICAL TRIAL: NCT03032016
Title: A Multi-centre, Multinational, Prospective Observational Registry to Collect Safety and Outcome Data in Patients Diagnosed With Severe Hepatic Veno-occlusive Disease (VOD) Following Hematopoietic Stem Cell Transplantation (HSCT) and Treated With Defitelio®
Brief Title: European VOD Registry
Status: Completed | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Other Study IDs: DF VOD-2013-03-REG
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Hepatic Veno-Occlusive Disease
Keywords: VOD; Defibrotide; Defitelio; Registry; SOS
MeSH Terms: conditions — Hepatic Veno-Occlusive Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sVOD patient treated with defibrotide: Patient diagnosed with severe hepatic VOD and treated with defibrotide

SUMMARY:
Following the licencing of a new drug, Defitelio®, indicated for the treatment of severe Veno-Occlusive Disease of the liver (sVOD), a rare but serious complication of haematopoietic stem cell transplantation (HSCT), as a specific obligation (SOB), the manufacture and marketing Authorisation Holder (MHA) (Gentium, a Jazz Pharmaceuticals Company) was required by PRAC (Pharmacovigilance Risk Assessment Committee) to set up a disease registry to collect safety and outcome data, and to assess patterns of utilization of Defitelio® in the post-approval setting. This registry is a Post Authorization Safety Study (PASS), is being coordinated in collaboration with the European Society for Blood and Marrow Transplantation (EBMT). For this study, anonymised clinical data are being collected from patients who develop VOD and and treated with and patients who have been treated with Defitelio® for conditions other than sVOD.

The study DOES NOT involve decisions about treatment, which are clinical decisions, but merely collection of data for patients who develop this complication, whether or not they receive treatment and for patients who are treated with Defitelio® for any other reasons.The study DOES NOT involve decisions about treatment, which are clinical decisions, but merely collection of data for patients who develop this complication, whether or not they receive treatment and for patients who are treated with Defitelio® for any other reasons.

DETAILED DESCRIPTION:
Defitelio® was granted a Marketing Authorisation in Europe under exceptional circumstances on 18 October 2013. Defitelio® is indicated for the treatment of severe hepatic Veno-Occlusive Disease (sVOD) also known as sinusoidal obstruction syndrome (SOS) in haematopoietic stem-cell transplantation (HSCT) therapy.

It is indicated in adults and in adolescents, children and infants over 1 month of age.

As required by the risk management plan, Gentium set up a disease registry to collect safety and outcome data, and to assess patterns of utilization of Defitelio® in the post-approval setting.

This is a multi-centre, multinational and prospective observational (non-interventional) disease registry of patients with severe hepatic VOD following HSCT and treated with Defitelio®.

The registry will be conducted in European transplant centres that are members of the European Society for Blood and Marrow Transplantation (EBMT).

The main objective of the registry is to assess the incidence rate of specific SAEs (Serious Adverse Events) of interest (including fatalities) in patients with severe hepatic VOD post-HSCT treated with Defitelio®.

Secondary objectives are:

* To describe the population treated with Defibrotide (age, gender, patients with pre-existing liver or severe renal insufficiency; patient with intrinsic lung disease)
* To determine the incidence rate of multiorgan failure (MOF) and Graft versus host disease (GvHD) in adult and paediatric patients receiving Defibrotide.
* To determine survival by Day+100 post-HSCT, overall mortality and mortality due to VOD in patients treated with Defibrotide.
* To determine the rate of VOD and VOD with MOF resolution any time after treatment initiation in patients treated with Defibrotide.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hematopoietic stem cell transplantation and diagnosed with severe hepatic VOD, who agree to participate in the study (Main population).
* Patients treated with defibrotide for another condition than severe hepatic VOD (Secondary population) in the scope of hematopoietic stem cell transplantation .

Exclusion Criteria:

* There will not be any specific exclusion criteria; however contraindications, special warnings and precautions for use as detailed in the SPC will have to be considered by the treating physician.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients will be selected by the treating physicians working in hospitals being part of the European society for Bone Marrow Transplantation network.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Incidence rate of specific SAE of interest | over 12 months
  Assess the incidence rate of specific SAEs of interest (including fatalities) in patients with severe hepatic VOD post-HSCT treated with Defitelio®

SECONDARY OUTCOMES:
Describe the population treated | Enrolment
  To describe the population treated with Defitelio® (age, gender, patients with pre-existing liver or severe renal insufficiency; patient with intrinsic lung disease)
GvHD incidence | over 12 months
  Determine the incidence rate of Graft versus host disease (GvHD) in adult and paediatric patients receiving Defitelio®
Survival | over 12 months
  To determine survival by Day+100 post-HSCT, overall mortality and mortality due to VOD in patients treated with Defitelio®
VOD/MOF Resolution | over 12 months
  To determine the rate of VOD and VOD with MOF resolution any time after treatment initiation in patients treated with Defitelio®

CONTACTS AND LOCATIONS:
Locations (53):
- France (22):
  - CHRU Angers, Maladies du Sang, Angers
  - CHU Bordeaux Groupe hospitalier Pellegrin Enfants, Bordeaux
  - CHU d'Estaing, Clermont-Ferrand
  - CHRU de Lille, Lille
  - Hôpital Jeanne de Flandre, Lille
  - CHRU Limoges, Limoges
  - IHOP, Lyon
  - Hôpital d'enfants de la Timone, Mare aux Daims
  - Institut Paoli Calmette, Marseille
  - CHU Lapeyronie, Montpellier
  - CHU Nantes, Nantes
  - Hôpital de l'ARCHET, Nice
  - Hôpital Saint Antoine, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Tenon, Paris
  - Institut Curie, Paris
  - Hôpital Haut Leveque, Pessac
  - Hôpital de la Miletrie, Poitiers
  - CHU Hautepierre, Strasbourg
  - IUTC Oncopole, Toulouse
  - Institut Gustave Roussy (Pediatrics), Villejuif
  - Institut Gustave Roussy, Villejuif
- Italy (19):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Ospedale di Careggi, Florence
  - UO Oncoematologia Ospedale Pediatrico Mayer, Florence
  - Institute G. Gaslini, Genova
  - Ospedale San Raffaele, Milan
  - Ospedale Ca' Granda Ospedale Maggiore di Milano, Milan
  - Ospedale di Niguarda Ca' Granda, Milan
  - Clinica di oncoematologia pediatrica, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale Santa Maria de la Misericorda, Perugia
  - Ospedale San Carlo, Potenza
  - IRRCS Ospedale Pediatrico Bambino Gesù, Roma
  - Universita Cattolica S. Cuore, Roma
  - La Sapienza University Hospital, Rome
  - AOU Citta della salute e delle Scienza, Torino
  - Ospedale Infantile Regina Margherita, Torino
  - Istituto per l'Infanzia IRCCS Burlo Garofolo, Trieste
  - Clinica Ematologica-Azienda Ospedaliero Universitaria, Udine
  - Policlinico G.B. Rossi, Clinica di Oncoematologia Pediatrica, Verona
- Inst. Portugues Oncologia o Lisboa, Lisbon, Portugal
- United Kingdom (11):
  - Birmingham Children's Hospital, Birmingham
  - Birmingham Heartlands Hospital, Birmingham
  - Bristol Royal Hospital for Children, Bristol
  - Great Ormond Street Hospital Children's Charity, London
  - Imperial College, London
  - St George's Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Great North Children's Hospital, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - John Radccliffe Children's Hospital, Oxford
  - Plymouth Hospitals NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mohty M, Battista ML, Blaise D, Calore E, Cesaro S, Maximova N, Perruccio K, Renard C, Wynn R, Zecca M, Labopin M, Hanvesakul R, Amber V, Ryan RJ, Lawson S, Ciceri F. A multicentre, multinational, prospective, observational registry study of defibrotide in patients diagnosed with veno-occlusive disease/sinusoidal obstruction syndrome after haematopoietic cell transplantation: an EBMT study. Bone Marrow Transplant. 2021 Oct;56(10):2454-2463. doi: 10.1038/s41409-021-01265-2. Epub 2021 May 31. PMID 34059801